CLINICAL TRIAL: NCT02314806
Title: Effect of Gentamicin Versus Clindamycin Versus Normal Saline Lavage of the Axillary Surgical Bed After Lymph Node Dissection on Drainage Discharge Volume
Brief Title: Gentamicin Versus Clindamycin Versus Normal Saline Lavage in Axilla
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Medicine Doctor, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HGUE 2014-12
Record Dates: First submitted 2014-12-07; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Therapeutic Irrigation; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Irrigation with Gentamicin solution (Experimental): The surgical bed is irrigated with a gentamicin solution
  Interventions: Drug: Irrigation with gentamicin solution
- Irrigation with Clindamycin solution (Experimental): The surgical bed is irrigated with a clindamycin solution
  Interventions: Drug: Irrigation with Clindamycin solution
- Irrigation with Normal saline (Placebo Comparator): The surgical bed is irrigated with normal saline
  Interventions: Drug: Irrigation with Normal saline

INTERVENTIONS:
Drug: Irrigation with gentamicin solution — The surgical bed is irrigated with a gentamicin solution
  Other Names: Irrigation of the surgical bed with gentamicin solution
  Arms: Irrigation with Gentamicin solution
Drug: Irrigation with Clindamycin solution — The surgical bed is irrigated with a clindamycin solution
  Other Names: Irrigation of the surgical bed with Clindamycin solution
  Arms: Irrigation with Clindamycin solution
Drug: Irrigation with Normal saline — The surgical bed is irrigated with normal saline
  Other Names: Irrigation of the surgical bed with normal saline
  Arms: Irrigation with Normal saline

SUMMARY:
The patients undergoing axillary lymph node dissection were randomized into 3 groups: patients undergoing lavages with normal saline (Group 1), patients undergoing lavage gentamicin solution (Group 2) and patients undergoing lavage with a clindamycin solution (Group 3). Drainage volume discharge is investigated

DETAILED DESCRIPTION:
The patients undergoing axillary lymph node dissection were randomized into 3 groups: patients undergoing 2 lavages with 500 ml normal saline (Group 1), patients first undergoing lavage with 500 ml normal saline followed by a second lavage with a 500 ml of a gentamicin (240 mg) solution (Group 2) and patients first undergoing lavage with 500 ml normal saline followed by a second lavage with 500ml of a clindamycin (600mg) solution (Group 3). Drainage volume discharge is investigated

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast neoplasms
* plans to undergo an elective ALND of Berg's levels I and II due to axillary metastasis determined preoperatively by core biopsy or evidence of metastasis in the SLNB in the intraoperative or in the differed analysis.

Exclusion Criteria:

* allergy to any of the antibiotic drugs used
* chronic renal failure due to possible toxicity of gentamicin
* patients undergoing a modified radical mastectomy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Drainage volume discharge | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, MD, PhD, Principal Investigator — Hospital General de Elche

REFERENCES:
- [Derived] Oller I, Ruiz-Tovar J, Cansado P, Zubiaga L, Calpena R. Effect of Lavage with Gentamicin vs. Clindamycin vs. Physiologic Saline on Drainage Discharge of the Axillary Surgical Bed after Lymph Node Dissection. Surg Infect (Larchmt). 2015 Dec;16(6):781-4. doi: 10.1089/sur.2015.020. Epub 2015 Aug 5. PMID 26244837